CLINICAL TRIAL: NCT02733835
Title: Novel Vital-sign Patient-assisted Intravenous Analgesia With Remifentanil for Labour Pain to Reduce Maternal Desaturation and Improve Analgesic Titration: a Prospective Cohort Study
Brief Title: VPIA Remifentanil for Labour Pain to Reduce Maternal Desaturation and Improve Analgesic Titration
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIRB/2015/2352
Record Dates: First submitted 2015-12-30; First posted 2016-04-12 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-01

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Remifentanil (Experimental): Remifentanil Patient Controlled Analgesia
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Vital signs-controlled, patient assisted intravenous analgesia using remifentanil
  Other Names: Ultiva

SUMMARY:
This study is a prospective cohort study aiming to evaluate an improved VPIA remifentanil algorithm which would benefit labouring mothers who are unable or unwilling to receive epidural analgesia

DETAILED DESCRIPTION:
This study trials a new Vital signs-controlled patient-assisted intravenous analgesia (VPIA) regimen using a purpose-built pump that aims to enhance the efficacy, safety and personalization of remifentanil therapy for labouring women. The system studies the parturient's pattern of analgesic use in 15 minute epochs and titrates the demand doses and basal infusion rate to maintain a plasma level of remifentanil that is appropriate for the degree of pain felt.

The system incorporates vital signs (pulse oximetry and heart rate values) into the algorithm which would temporarily stop the pump and step down doses accordingly when predefined critical values are reached.

ELIGIBILITY:
Inclusion Criteria:

* Patients who choose to use parenteral opioid for pain relief with informed consent
* Patients who refuse labour epidural analgesia or with contraindication to epidural analgesia (eg. thrombocytopaenia, previous thoraco-lumbar spinal instrumentation)
* Gestational age of >= 36 weeks

Exclusion Criteria:

* Patients who are unable to understand instructions given regarding the use of patient controlled analgesia (PCA) or unable to self administer PCA boluses
* Patients with difficulty in communication due to language differences
* Patients with known hypersensitivity to remifentanil or any component of its formulation or to other fentanyl analogue
* Patients with severe respiratory disease
* Patients with history of drug dependence of recreational drug abuse
* Patients with unmanaged foetal bradycardia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Maternal desaturation | Duration of labour

SECONDARY OUTCOMES:
Maternal bradycardia | Duration of labour, an expected average of 24 hours
Apnoea/hypopnoea | Duration of labour, an expected average of 24 hours

OTHER OUTCOMES:
Side effects: pruritus | Duration of labour, an expected average of 24 hours
  Pruritus
Side effects: nausea vomiting | Duration of labour, an expected average of 24 hours
  Nausea/vomiting
Side effects: sedation | Duration of labour, an expected average of 24 hours
  Sedation
Maternal outcomes: duration of labour | Duration of labour, an expected average of 24 hours
  Duration of labour (minutes)
Maternal outcomes: duration of second stage | At delivery, an expected average of 1 hour
  Duration of second stage (minutes)
Maternal outcomes: pain score | Duration of labour, an expected average of 24 hours
  Maternal pain score (out of 10)
Maternal outcomes: satisfaction score | Duration of labour, an expected average of 24 hours
  Maternal satisfaction score (%)
Neonatal outcomes: birth weight | Immediately after birth
  Birth weight in grams
Neonatal outcomes: APGAR | Immediately after birth
  APGAR scores
Neonatal outcomes: cord blood pH | Immediately after birth
  Umbilical cord blood pH

CONTACTS AND LOCATIONS:
Overall Officials: Wan Ling Leong, MBBS FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No